CLINICAL TRIAL: NCT04648397
Title: The Effect of Chewing Duration on Blood Glucose Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Principal investigator, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NL74340.081.20
Record Dates: First submitted 2020-11-05; First posted 2020-12-01 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Glucose, High Blood; Glucose, Low Blood
Keywords: Chewing behaviour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short chewing (Experimental): Subjects consume two starch-based foods varying in fibre content e.g. brown rice and chick-peas in duplicate following a short chewing protocol.
  Interventions: Other: Low glycaemic load, high fibrous product; Other: High glycaemic load, low fibrous product
- Long chewing (Experimental): Subjects will consume two starch-based foods varying in fibre content e.g. brown rice and chick-peas in duplicate following a long chewing protocol.
  Interventions: Other: Low glycaemic load, high fibrous product; Other: High glycaemic load, low fibrous product

INTERVENTIONS:
Other: Low glycaemic load, high fibrous product — Test-lunch of 370 grams of chickpeas, seasoned with a herb- and spice mix to increase palatability. Glycaemic load 18.5. Consumed in duplicate.
Other: High glycaemic load, low fibrous product — Test-lunch of 257 grams of brown rice, seasoned with rice-oil and a herb- and spice mix to increase palatability. Glycaemic load 44.9. Consumed in duplicate.

SUMMARY:
This study aims to assess the impact of speed of consumption of two starch-based foods varying in fibre content on blood glucose levels in normal healthy subjects. Furthermore, the mediating roles of salivary amylase and particle size on blood glucose levels will be studied. The study has a randomized cross-over design. Subjects consume two test-lunches (chick peas and brown rice) in duplicate on 8 different test days, at either long or short chewing duration. Glucose responses will be monitored via a continuous glucose monitoring device and expectorated boluses will be collected during each test day for assessments of amylase activity and food particle size.

DETAILED DESCRIPTION:
Research suggests that high glucose level variability and large dips in glucose levels may have a negative impact on cognitive function and self-reported wellbeing. The way food is consumed (e.g. chewing duration) may regulate blood glucose levels. The underlying mechanism that links consumption speed to metabolic responses, satiation and health is largely unknown.

This study aims to assess the impact of speed of consumption of two starch-based foods varying in fibre content, on blood glucose levels in normal healthy subjects. Furthermore, the mediating roles of salivary amylase and particle size on blood glucose levels are studied.

The study has a randomized cross-over design. Each subject consumes two different test-lunches (chick peas and brown rice) in duplicate at either long or short duration. Their breakfast will be standardized during these 8 test days. For a duration of 12 days, blood glucose levels will be monitored via a continuous glucose device. Furthermore expectorated boluses will be collected for assessment of amylase activity and food particle size.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women (based on questionnaire, self-reported)
* Aged between 18 - 55 yrs
* BMI between 18.5 - 30 kg/m2
* In possession of a Smartphone running on iOS or Android

Exclusion Criteria:

* Diagnosed with Diabetes mellitus type 1 or 2
* Under treatment for neurological or psychiatric complaints, including eating disorders
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* Use of medication/supplements that may influence the study results, such as medicines known to interfere with glucose homeostasis. This will be judged by our medical doctor
* Following a diet or gained/lost >=5kg weight in the previous month.
* Coeliac disease or gluten intolerance
* Skin allergy, eczema or known sensitivity for plasters
* use of drugs
* Current smokers
* Using > 14 glasses of alcohol per week
* Having a food allergy for the test foods
* Participation in another clinical trial at the same time
* Suffering from a stomach emptying disorder
* Employed by or an intern at the FHCR group of Wageningen Food & Biobased Research.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Blood glucose responses in the 3 hrs following lunch | 12 days in total to cover all test days
  measured by a continuous glucose monitoring device

SECONDARY OUTCOMES:
Particle size of food bolus | on 4 of the 8 test days, at day 1, day 2, day 3 and day 4 or day 5, day 6, day 7 and day 8 depending on group
  measured in food boli of the test-lunches by image analysis
Amylase activity | at day 1
  measured in saliva
In vitro starch digestion rates in food bolus | on 4 of the 8 test days, at day 1, day 2, day 3 and day 4 or day 5, day 6, day 7 and day 8 depending on group
  assessed in food boli of the test-lunches by making use of INFOGEST 2.0 protocol

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Stieger M, Capuano E, Forde CG, van der Haar S, Ummels M, van den Bosch H, de Wijk R. Influence of oral processing behaviour and bolus properties of brown rice and chickpeas on in vitro starch digestion and postprandial glycaemic response. Eur J Nutr. 2022 Dec;61(8):3961-3974. doi: 10.1007/s00394-022-02935-7. Epub 2022 Jun 30. PMID 35773354